CLINICAL TRIAL: NCT05113511
Title: A Randomized, Double-blind, Parallel-controlled Phase I Clinical Study Comparing the Pharmacokinetics, Safety and Immunogenicity of SCT510 With Bevacizumab (Avastin®) in Chinese Healthy Males
Brief Title: PK and Safety of SCT510
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Sinocelltech Ltd. (Industry)
Responsible Party: Principal Investigator, shentu jianzhong, Ph.D.(Pharm）, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCT510NSCLC01
Record Dates: First submitted 2021-11-08; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: pharmacokinetics; immunogenicity; biosimilar; phase I; anti-VEGF monoclonal antibody
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT510 (Experimental): SCT510
  Interventions: Drug: SCT510
- bevacizumab (Active Comparator): bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: SCT510 — Subjects received a single intravenous infusion (3 mg/kg) of SCT510 for 90 minutes , and the volume of administration was calculated based on the subject's weight.
  Arms: SCT510
Drug: Bevacizumab — Subjects received a single intravenous infusion (3 mg/kg) of bevacizumab for 90 minutes , and the volume of administration was calculated based on the subject's weight.
  Arms: bevacizumab

SUMMARY:
This is a randomized, double-blind, parallel-controlled phase I clinical study comparing the pharmacokinetics, safety and immunogenicity of SCT510 with bevacizumab (Avastin®) in Chinese healthy males.

DETAILED DESCRIPTION:
Eighty-four subjects randomly (1:1) received a 3 mg/kg dose of SCT510 or bevacizumab infusion for 90 min and followed up for 99 days. The screening period of this study is 14 days. Subjects will be admitted to the research center on day-1 and will be allowed to leave the research center with relevant observation and evaluation on day 5 (96 hours) after the completion of the administration. Subjects were asked to return for 10 follow-up visits respectively according to this research protocol, on the day 8, day 15, day 22, day 29, day 43, day 57, day 64, day 71, day 85 and day 99.

All subjects in each group will be blinded after blood/urine collection and safety evaluation.

Blood samples will be tested by a validated LC/MS method for pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who fully understand the purpose, content, benefits and possible adverse reactions of the test and voluntarily sign written informed consent prior to the commencement of any test-related activities.
2. Healthy males, aged 18 to 45 years (including 18 and 45 years).
3. Male subjects weighed 45-100 kg (including 45 and 100 kg), body mass index (BMI) was 19.0-25.0 kg/m2 (including 19.0 and 25.0 kg/m2), where BMI = body weight (kg)/height2 (m2).
4. The subject agrees to use reliable contraceptive methods (such as abstinence, sterilization, birth control pills, injectable contraceptive meprogesterone or subcutaneous implantation) for himself and his partner during the study period and for 6 months after the infusion of study drugs.

Exclusion Criteria:

1. History of hypertension or abnormal blood pressure at screening/baseline [SBP >140 mmHg and/or diastolic blood pressure >90 mmHg confirmed by one repeat measurement on the same day];
2. Clinically significant proteinuria examination or history of proteinuria assessed by the investigator;
3. Abnormal physical examination or examination results (e.g., chest X-ray, laboratory examination) are considered clinically significant by the investigator;
4. Have received any antibody or protein drug or small molecule targeted drug therapy targeting VEGF or VEGF receptor in the past 1 year;
5. Use of any biological product or live viral vaccine within 3 months prior to drug infusion, or use of any monoclonal antibody within 12 months;
6. Have hereditary bleeding tendency or coagulopathy, or have a history of thrombosis or bleeding;
7. History of digestive tract perforation or fistula;
8. Unhealed wounds, ulcers or fractures, or those who had undergone major surgery within the previous 2 months or were expected to undergo major surgery within the study period or 2 months after the end of the study;
9. Use a prescription or over-the-counter drug or nutraceutical product within the 5 half-life of the drug or nutraceutical product or within 2 weeks prior to use of the study drug, whichever is longer. Herbal supplements should be discontinued 28 days prior to use of the study drug;
10. Hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody test positive;
11. Known allergy to bevacizumab or any of its excipients;
12. Known history of allergic diseases or allergies;
13. People with a history of severe allergy, allergy to protein products, rat-derived products and related ingredients of experimental drugs;
14. Blood donation history within 3 months prior to drug infusion;
15. Has received any other investigational drug treatment or participated in another interventional clinical trial within 3 months prior to screening;
16. History of alcohol or drug abuse in the 12 months prior to screening; Subjects were unable to abstain from alcohol within 72 hours prior to administration and throughout the trial;
17. A history of mental illness;
18. Have pregnancy plans during the trial ;
19. Unable to complete the study according to protocol requirements during the study;
20. Conditions considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336, 504，672, 1,008, 1,344, 1,512, 1,680, and 2,016 hours after SOI ]
  area under the concentration-time curve from time zero (pre-dose) extrapolate area under the concentration-time curve from time zero (pre-dose) extrapolated to infinity
AUC0-last | pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336, 504，672, 1,008, 1,344, 1,512, 1,680, and 2,016 hours after SOI ]
  area under the concentration-time curve from time zero (pre-dose) extrapolated to last quantifiable concentration (AUC0-t)
Cmax | pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336, 504，672, 1,008, 1,344, 1,512, 1,680, and 2,016 hours after SOI ]
  Maximum Serum Concentration

SECONDARY OUTCOMES:
Tmax | pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336, 504，672, 1,008, 1,344, 1,512, 1,680, and 2,016 hours after SOI ]
  Time to Cmax
Number of Participants With Anti-Drug Antibody Positive | up to 99 days
  number of participants with anti-drug antibody positive at post-dose
Number of Participants With neutralizing antibody Positive | up to 99 days
  number of participants with neutralizing antibody positive at post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong Q, Jiao Y, Li D, Ma H, Wu K, Xie L. Population Pharmacokinetics of SCT510 (a Bevacizumab Biosimilar) and Avastin(R) in Healthy Subjects and Patients with Non-squamous Non-small Cell Lung Cancer. Clin Drug Investig. 2026 Feb;46(2):143-157. doi: 10.1007/s40261-025-01518-8. Epub 2026 Jan 6. PMID 41495391
- [Derived] Wu J, Wu G, Xie L, Lv D, Xu C, Zhou H, Wu L, Zhang J, Shentu J. A Randomized, Double-Blind, Parallel-Controlled Phase I Study Comparing the Pharmacokinetics, Safety, and Immunogenicity of SCT510 to Bevacizumab (Avastin(R)) in Healthy Chinese Males. Drugs R D. 2023 Jun;23(2):175-183. doi: 10.1007/s40268-023-00424-8. Epub 2023 May 29. PMID 37247166